CLINICAL TRIAL: NCT02363075
Title: A Study Evaluating Dexamfetamine Sulphate in Patients With Glioma Suffering From Severe Asthenia. A Phase III Double-blind Randomized Placebo-controlled Trial
Brief Title: Dexamfetamine Sulphate in Patients With Glioma Suffering From Severe Asthenia
Acronym: DXA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P110501
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Glioma
Keywords: dexamfetamine sulphate; severe asthenia; glioma; MFI-20; double-blind; stabilisation phase
MeSH Terms: conditions — Glioma; Asthenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamfetamine sulphate (Experimental): Dexamfetamine Sulphate 5 mg Tablets
  Interventions: Drug: Dexamfetamine sulphate
- placebo (Placebo Comparator): Aspect tablets identical to the active
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexamfetamine sulphate — 10mg/day per os for the first ten days, 20mg/day for the ten following days, 30mg/day until D90.
  Arms: Dexamfetamine sulphate
Drug: placebo — 10mg/day per os for the first ten days, 20mg/day for the ten following days, 30mg/day until D90.
  Arms: placebo

SUMMARY:
The main purpose of this study is to estimate the efficiency at 3 months of dexamfetamine sulphate on the MFI 20 scale in severe fatigue of patients with stabilized gliomas.

DETAILED DESCRIPTION:
Quality of life of patients with stabilized gliomas is often impacted by a severe physical and psychological fatigue resulting from both tumor and side effects of treatments.

It is a randomized double blind Placebo-Controlled Trial evaluating the effect of dexamfetamine sulphate on severe fatigue in glioma patients. Half of the participants will receive dexamfetamine sulphate and the other half will receive a placebo. Neither the participant nor the study doctor will know what group they are in.

The main objective is to assess the impact at 3 months of dexamfetamine sulphate in patients suffering from a RANO stable or responsive glioma complaining of a severe fatigue (quantified by the Multidimensional Fatigue inventory - MFI 20 scale).

The secondary objectives include: evaluation of side effects, quality of life, cognitive functions, depression, variation in time of both fatigue scales MFI 20 and VAS.

58 patients will be included. In patients complaining of severe asthenia, with a non progressive neuro-oncological disease, and without criteria of depression revealed by HAD (Hospital Anxiety and Depression) scale, evaluation of fatigue will be done with the MFI 20 scale. Patients with a MFI 20 score ≥60/100 and corresponding to inclusion criteria will be invited to participate.

After randomisation, a baseline evaluation will be done, including MFI20, Norris VAS, EORTC QLQ-C30, Mattis scale, Trail Making Test, Grober and Buschke, Wisconsin Card Sorting Test , HAD scale and Marin scale.

Patients will receive, in a double blinded way, six pills a day either of dexamphetamine sulfate (15 mg*2) or of placebo, during 3 months, after an initial phase of progressive increasing levels of dose every 10 days, depending on tolerance.

The evaluation of fatigue, quality of life will be done every month during the 3 months of treatment. The cognitive evaluation will be done at 3 months.

The main criteria of evaluation is the variation during 3 months of the MFI 20 score in non progressive patients.

ELIGIBILITY:
Inclusion criteria :

* Patients complaining of a severe asthenia defined as a MFI 20 score ≥ 60/100
* Patients suffering from histologically proven gliomas
* Patients with responsive or stable disease (according to RANO criteria) for at least 3 months, either still on chemotherapy or only being under simple surveillance
* stable dosage of steroids for at least 1 week
* Time elapsed post-radiotherapy more than 3 months
* HAD score of depression ≤8
* Karnofsky performance index ≥ 60
* ≥ 18 years of age
* contraceptive measures
* written informed consent
* Depending from the french system of health assurance

Exclusion criteria :

* Severe aphasia or other symptoms compromising the tests execution
* concomitant uncontrolled pathology
* Known symptomatic or constitutional cardiovascular disease, (cardiac arrhythmia, recent myocardial infarction, chest pain, history of unstable angina) and/or uncontrolled hypertension, (≥ 16/10), arteriosclerosis, cardiac abnormality detected at the initial cardiac echography.
* Hyperthyroidism
* Known hypersensitivity to dexamphetamine or related compounds
* Glaucoma
* Porphyria
* Hemoglobin level of less than 10,0 g/dL
* Alcohol or drug abuse,
* Agitation
* Tourette's syndrome
* Patients who have been receiving MAO inhibitors during the past 14 days
* Hereditary hypersensitivity to galactose, Lapp lactase deficiency or glucose-galactose malabsorption syndrome
* Hereditary hypersensitivity to saccharose, glucose-galactose malabsorption syndrome or saccharase-isomaltase deficiency
* Pregnant or lactating woman
* Non french speaker
* History of psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-07 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue inventory - MFI 20 scale score | 3 months
  improvement of the MFI 20 score between the inclusion and the evaluation at 3 months in case of non progressive disease during this period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Florence LAIGLE-DONADEY, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitie Salpetriere, Paris, France